CLINICAL TRIAL: NCT05984108
Title: Clinical, Radiological, Histological and Molecular Features of a Cohort of Melanocytic Tumors of the Central Nervous System
Brief Title: Clinical, Radiological, Histologic and Molecular Features of a Cohort of Melanocytic Tumors of the Central Nervous System
Acronym: MelaMen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Guillaume GAUCHOTTE, PhD, Central Hospital, Nancy, France
Other Study IDs: 2022PI132
Record Dates: First submitted 2023-06-25; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-07

CONDITIONS: Meningeal Melanocytoma; Meningeal Melanomatosis; Meningeal Melanocytosis; Meningeal Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Formalin-fixed Paraffin-embedded tumor samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Meningeal melanocytoma
- Meningeal melanoma
- Meningeal melanomatosis
- Meningeal melanocytosis

SUMMARY:
Primary melanocytic tumors of the central nervous system are rare lesions and occur develop from leptomeningeal melanocytes. The WHO classification of tumors of the central nervous system in its most recent version (2021) distinguishes on the one hand the circumscribed melanocytic tumors including melanocytoma, benign, and its slope malignant, meningeal melanoma, with an intermediate grade lesion in between, called intermediate grade melanocytoma. They are to be distinguished from diffuse tumors or multifocal diseases such as melanocytosis and its malignant corollary, melanomatosis. The main current challenge is to distinguish them from their differential diagnoses, namely metastasis of a cutaneous or extrac-cutaneous melanoma mainly and on the other hand other pigmented entities occuring in the CNS such as malignant melanic tumor of the peripheral nerve sheath (MMNST, formerly "melanotic schwannoma").

DETAILED DESCRIPTION:
The discovery within the CNS of a tumor of melanocytic nature requires the realization an exhaustive assessment (dermatological examination, whole body imaging), especially in the event of signs histological evidence of malignancy (marked atypia, mitoses, infiltration of the parenchyma), in order to look for unnoticed cutaneous melanoma. In the absence of primary lesion found outside the nervous system, the question of a primary lesion with a meningeal starting point arises. A molecular characterization is then required, in order to highlight mutations recurrent spores of the GNA11 or GNAQ genes, classically not found in the cutaneous melanomas, the latter presenting different genetic alterations (BRAF, NRAS, KIT etc). Other rarer alterations such as PLCB4 or CYSLTR2 are also described in these meningeal melanocytic tumors, but are not part of the gene panels of routine. On the other hand, the discovery of a circumscribed melanocytic lesion, in particular intradural extramedullary and spindle cells, should suggest the differential diagnosis malignant melanotic nerve sheath tumor (MMNST, malignant melanotic nerve sheath tumor), formerly called "melanotic schwannoma". Distinguish them histologically can be tricky. This differential diagnosis is important, the MMNST entering often in the context of Carney syndrome, of autosomal dominant transmission, responsible for other conditions requiring multidisciplinary follow-up (cardiac myxoma, endocrine disorders). Recent advances in molecular biology have opened up new possibilities for the diagnosis and classification of brain tumours. One of them is the methylome, studying the epigenetic signature of a tumor via its methylation profile.

These epigenetic modifications play an important role in regulating the expression genes and are now well known to be involved in the development and cancer progression. This tool has been integrated into the new WHO 2021 classification of CNS tumors and constitutes for certain entities an essential criterion for their diagnosis final. The publication by Capper et al. in 2018, entitled "DNA methylation-based classification of central nervous system tumours" illustrates this point. It was highlighted that meningeal melanocytic tumors cluster separately from other types of tumors, including cutaneous melanomas. Three methylation classes exist currently in version 12.5 of the classifier developed by the University of Heidelberg (www.molecularneuropathology.com): a class of methylation specific to the metastases of melanoma, one for malignant melanotic peripheral nerve sheath tumors, and a titled melanocytoma (which includes entities with similar profiles: melanocytoma and meningeal melanoma but also uveal melanoma). He does not exist to date of methylation class for diffuse meningeal melanocytic tumors(melanocytosis and its malignant corollary melanomatosis).

To conclude, meningeal melanocytic tumors are a group of tumors of the system central nervous system rare but for which it is necessary to make a diagnosis of certainty The WHO classification proposed in 2021 is based on an integrative histo-molecular approach, but for which the community medicine still lacks perspective. In particular, when using this new classification, it there are difficulties in classifying certain tumours, presenting clinical aspects, discordant radiological, histopathological and molecular findings.

The aims of this study are therefore to classify melanocytic tumors according to the new WHO 2021 classification of central nervous system tumors, to describe their clinical, radiological, histological and molecular characteristics, to define new prognostic criteria (mitotic index, Ki-67 , immunohistochemical markers such as BAP1 and p16) and to establish clinico-radio-histo-molecular correlations.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a primitive meningeal melanocytic tumor

Exclusion Criteria:

* Patient with metastatic extrameningeal melanoma

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primitive meningeal melanocytic tumors
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Diagnosis according to WHO classification of CNS tumors (5th edition) | at baseline (initial report)
  Histologic diagnosis according to WHO classification of CNS tumors (5th edition) among these 5 options : melanocytoma, intermediate-grade melanocytoma, melanoma, melanocytosis, melanomatosis
Mitotic index | at baseline (initial report)
  Number of mitoses per square millimetre
Age | At baseline
  Age in years
Sex | At baseline
  Male or female
Ki-67 | At time of initial diagnosis
  Proliferation index Ki-67, assessed by immunohistochemistry, counted on 500 cells
T1-weighted sequence signal | At time of initial diagnosis
  Radiologic feature : tumor T1-weighted sequence signal on MRI (hyposignal, isosignal, hypersignal)
Enhancement after gadolinium injection | At time of initial diagnosis
  Radiologic feature: tumor enhancement after gadolinium injection on MRI

SECONDARY OUTCOMES:
Overall survival | From date of initial diagnosis until the date of death of any cause assessed up to 10 years
  Time from diagnosis to death
Progression-free survival | From date of initial diagnosis until the date of first documented progression assessed up to 10 years
  Time from diagnosis to first progression

CONTACTS AND LOCATIONS:
Locations (1):
- Nancy University Hospital Center, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Koelsche C, Hovestadt V, Jones DT, Capper D, Sturm D, Sahm F, Schrimpf D, Adeberg S, Bohmer K, Hagenlocher C, Mechtersheimer G, Kohlhof P, Muhleisen H, Beschorner R, Hartmann C, Braczynski AK, Mittelbronn M, Buslei R, Becker A, Grote A, Urbach H, Staszewski O, Prinz M, Hewer E, Pfister SM, von Deimling A, Reuss DE. Melanotic tumors of the nervous system are characterized by distinct mutational, chromosomal and epigenomic profiles. Brain Pathol. 2015 Mar;25(2):202-8. doi: 10.1111/bpa.12228. Epub 2014 Dec 15. PMID 25399693
- [Background] Kusters-Vandevelde HV, Kusters B, van Engen-van Grunsven AC, Groenen PJ, Wesseling P, Blokx WA. Primary melanocytic tumors of the central nervous system: a review with focus on molecular aspects. Brain Pathol. 2015 Mar;25(2):209-26. doi: 10.1111/bpa.12241. PMID 25534128
- [Background] Griewank KG, Koelsche C, van de Nes JAP, Schrimpf D, Gessi M, Moller I, Sucker A, Scolyer RA, Buckland ME, Murali R, Pietsch T, von Deimling A, Schadendorf D. Integrated Genomic Classification of Melanocytic Tumors of the Central Nervous System Using Mutation Analysis, Copy Number Alterations, and DNA Methylation Profiling. Clin Cancer Res. 2018 Sep 15;24(18):4494-4504. doi: 10.1158/1078-0432.CCR-18-0763. Epub 2018 Jun 11. PMID 29891723